CLINICAL TRIAL: NCT07221058
Title: Adaptive Radiation BOost for Rectal Cancer: a Phase I Dose Escalation Study (ARBOR)
Brief Title: Adaptive Radiation Boost for Rectal Cancer
Acronym: ARBOR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT-231; 25-1024 (Other: FCCC IRB)
Record Dates: First submitted 2025-10-22; First posted 2025-10-27 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Rectum Cancer, Adenocarcinoma
Keywords: Adaptive Radiation Therapy; Rectum Cancer; Adenocarcinoma; Organ Preservation; Total Mesorectal Excision
MeSH Terms: conditions — Rectal Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adaptive Radiotherapy Boost Following Standard Pelvic Chemoradiation (Experimental): Adaptive Radiotherapy
  Interventions: Radiation: Adaptive Radiotherapy Boost

INTERVENTIONS:
Radiation: Adaptive Radiotherapy Boost — Patients will receive one boost fraction every two weeks, targeting the primary tumor within the rectum plus a 2 mm Planning Target Volume (PTV) margin. Any regional lymph nodes that measure at least 5 mm in short axis on the day of treatment will receive treatment with the ART dose being given to the primary rectal tumor.

SUMMARY:
The goal of this clinical trial is to find out if giving extra adaptive radiation therapy after standard chemoradiation treatment is safe and helpful for people with rectal cancer.

The main questions the study aims to answer are:

* Can this approach help target the most aggressive cancer cells more accurately, while protecting nearby healthy tissue?
* Can it reduce the side effects that people may experience during treatment?

Participants will:

* First receive standard treatment: radiation (45 Gy in 25 sessions) along with a chemotherapy pill called capecitabine.
* Then get extra radiation using MRI scans every two weeks to adjust the treatment based on how the tumor responds.
* Use a small balloon during treatment to help aim the radiation and protect healthy areas.
* Finally, receive additional chemotherapy (such as FOLFOX) for four months.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically or cytologically confirmed rectal adenocarcinoma.
2. Subjects must have T2-3, N0-1, M0 rectal cancer. Staging will be done by MRI pelvis and CT chest and abdomen with contrast. PET-CT will be an acceptable alternative for the CT chest and abdomen.
3. Subjects must be willing to undergo MRI scans.
4. Age ≥18 years.
5. ECOG performance status 0 or 1.
6. Estimated survival of ≥ 12 months.
7. Subjects must have normal organ and marrow function as defined below

   * Absolute neutrophil count > =1,000/mcL
   * Platelets >= 75,000/mcL
   * Total bilirubin < 3 mg/dL
8. Subjects must be able to tolerate the chemotherapy regimens outlined in the treatment plan (Section 5.0), both before and after ART.

   * Before ART: Capecitabine at a dose of 825 mg/m²
   * After ART: FOLFOX combination chemotherapy, or 5-FU, or capecitabine
9. Subjects must possess the ability to understand and willingness to sign a written informed consent and HIPAA consent document. Translation services including translation of informed consent documents will be provided, as feasible, to encourage diversity of inclusion of eligible patients.

Exclusion Criteria:

1. Subjects who have been previously treated for rectal cancer are excluded.
2. Subjects with rectal cancer involving the anal canal are excluded. (Rectal cancer abutting the anal canal will be allowed.)
3. Subjects must not be receiving any other investigational agents.
4. Subjects may not have had prior pelvic radiation.
5. Subjects should not have had a cancer actively treated within the last 3 years, excluding non-melanoma skin cancer.
6. Subjects must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Any condition or significant co-morbidity that prevents safe delivery of ART per the discretion of the treating physician(s).
8. Subjects must not be pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
MTD will be evaluated by monitoring the rate of dose limiting toxicities (DLTs) defined as acute Grade 2+ gastrointestinal toxicity probably or definitely related to radiation. | From the initiation of rectal adaptive radiotherapy boost to 90 days after the last dose of boost, for a total of ~ 120 days.
Feasibility of a rectal boost that targets at least 90% of the rectal planning tumor volume with the 80% prescribed dose while limiting the outer 3 mm of the rectal wall to no more than 50% of the prescription dose delivered to 0.1cc. | From the ART boost initiation to the end of the ART boost, for a period of ~ 5 weeks
  Feasibility will be determined based on successful implementation and completion of standard chemoradiotherapy followed by experimental rectal adaptive radiotherapy boost utilizing CT-MR fusion that targets at least 90% of the rectal PTV_Eval with the 80% prescribed dose while limiting the outer 3 mm of the rectal wall to no more than 50% of the prescription dose delivered to 0.1cc in ≥ 70% of ART fractions for the patient population enrolled in the study. This will be assessed at the MTD.

SECONDARY OUTCOMES:
Estimate the efficacy of bi-weekly adaptive radiotherapy boost fractions by complete response rate, near complete response rate, and incomplete response rate as per Memorial Sloan Kettering Cancer Center (MSKCC) criteria. | From the end of rectal adaptive radiotherapy boost to the end of study, for a total of ~ 5 years.
Estimate total mesorectal excision (TME) free survival following treatment with the study regimen. | From the end of treatment to the end of the study, for a total of up to 5 years.
Estimate overall survival (OS) following treatment with the study regimen. | From the end of treatment to the end of study, for a total of up to 5 years.
Estimate early and late toxicity following treatment with the study regimen. | From the initiation of rectal radiation boost treatment to the end of the study, for a total of ~ 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Meyer, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States